CLINICAL TRIAL: NCT06437873
Title: Long-term Survival Outcomes of Total Thyroidectomy and Radioactive Iodine Therapy in Unilateral T3/T4 Follicular Thyroid Carcinoma:A Retrospective Propensity Score-Matched Study
Brief Title: Long-term Survival Outcomes of Total Thyroidectomy and Radioactive Iodine Therapy in Unilateral T3/T4 FTC
Status: Completed | Type: Observational
Sponsor: Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: DezhouH_2024_001
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Follicular Thyroid Cancer; SEER Database Analysis
Keywords: Retrospective analysis, follicular thyroid carcinoma, total thyroidectomy, long-term survival outcomes.
MeSH Terms: conditions — Adenocarcinoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Total Thyroidectomy (TT) Group: Patients with T3 or T4 stage follicular thyroid carcinoma who underwent total thyroidectomy
  Interventions: Procedure: Total Thyroidectomy (TT)
- No Total Thyroidectomy (No-TT) Group: Patients with T3 or T4 stage follicular thyroid carcinoma who did not undergo total thyroidectomy.
- Radioactive Iodine Therapy (RAIT) Group: Patients in the No-TT group who received radioactive iodine therapy.
  Interventions: Radiation: Radioactive iodine treatment(RAIT)
- No Radioactive Iodine Therapy (No-RAIT) Group: Patients in the No-TT group who did not receive radioactive iodine therapy.

INTERVENTIONS:
Procedure: Total Thyroidectomy (TT) — TT:Surgical removal of the entire thyroid gland.
  Groups: Total Thyroidectomy (TT) Group
Radiation: Radioactive iodine treatment(RAIT) — RAIT:Administration of radioactive iodine to eliminate remaining thyroid tissue or cancer cells.
  Groups: Radioactive Iodine Therapy (RAIT) Group

SUMMARY:
This study aims to thoroughly examine survival disparities in patients with T3 or T4 stage follicular thyroid carcinoma (FTC) as classified by the AJCC staging system. It compares outcomes between those who underwent total thyroidectomy (TT) and those who did not, and assesses the influence of radioactive iodine therapy (RAIT) on the survival of patients without TT. Utilizing the SEER database, a retrospective study identified patients diagnosed with T3 or T4 FTC, categorizing them into two cohorts: those treated with TT and those who were not (No-TT). The No-TT group was further analyzed to determine the impact of RAIT on patient survival. Propensity score matching (PSM) was applied to adjust for confounding variables. Survival analysis, including Kaplan-Meier survival curves and Landmark analysis, was conducted to evaluate the effects of surgical intervention and RAIT on overall survival (OS) and cancer-specific survival (CSS).

ELIGIBILITY:
Inclusion Criteria:1.The primary site code C73.9, denoting the thyroid gland;2.The International Classification of Diseases for Oncology, Third Edition (ICD-O-3) histology types comprising 8330 (Follicular adenocarcinoma, NOS), 8331 (Follicular adenocarcinoma well differentiated), 8332 (Follicular adenocarcinoma trabecular), 8335 (Follicular carcinoma, minimally invasive), and 8339 (Follicular thyroid carcinoma (FTC), encapsulated angioinvasive).

Exclusion Criteria:(1). Absence of T stage information or designation as T1, T2; (2). Missing surgery codes; (3). Cases not verified by histopathological analysis; (4). FTC not being the initial malignancy diagnosed in the patient; (5). Unknown survival duration or survival less than one month; (6). Presence of bilateral tumors.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The SEER database was established in 1973, serves as a public database and research resource developed by the National Cancer Institute (NCI) of the United States. It encompasses data covering approximately 30% of the U.S. population. The dataset for this retrospective study was obtained from the SEER Research Data, encompassing information from 17 registries as of November 2022, which includes cases recorded between the years 2000 and 2020.
Sampling Method: Probability Sample
Enrollment: 2957 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 10 years post-diagnosis
  Time from diagnosis until death from any cause.
Cancer-Specific Survival (CSS) | Up to 10 years post-diagnosis
  Time from diagnosis to death specifically from follicular thyroid carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Study Director — Dezhou Hospital Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with researchers upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 6 months after publication of the main study results and will be accessible for a period of 5 years.
Access Criteria: Researchers seeking access to the IPD must submit a methodologically sound proposal. Requests should be directed to the principal investigator and will be evaluated on the basis of scientific merit and ethical considerations.

REFERENCES:
- [Background] Daniels GH. Follicular Thyroid Carcinoma: A Perspective. Thyroid. 2018 Oct;28(10):1229-1242. doi: 10.1089/thy.2018.0306. Epub 2018 Aug 21. No abstract available. PMID 30039751
- [Background] Barbesino G, Goldfarb M, Parangi S, Yang J, Ross DS, Daniels GH. Thyroid lobe ablation with radioactive iodine as an alternative to completion thyroidectomy after hemithyroidectomy in patients with follicular thyroid carcinoma: long-term follow-up. Thyroid. 2012 Apr;22(4):369-76. doi: 10.1089/thy.2011.0198. Epub 2012 Mar 2. PMID 22385290
- [Background] Bal C, Satapathy S, Tupalli A, Ballal S. Propensity Score Matched Outcome Analysis of Lobar Ablation Versus Completion Thyroidectomy in Low-Risk Differentiated Thyroid Cancer Patients: Median Follow-Up of 11 Years. Thyroid. 2022 Oct;32(10):1220-1228. doi: 10.1089/thy.2022.0234. Epub 2022 Sep 22. PMID 35983596
- [Background] Choi JB, Lee SG, Kim MJ, Kim TH, Ban EJ, Lee CR, Lee J, Kang SW, Jeong JJ, Nam KH, Chung WY, Park CS. Oncologic outcomes in patients with 1-cm to 4-cm differentiated thyroid carcinoma according to extent of thyroidectomy. Head Neck. 2019 Jan;41(1):56-63. doi: 10.1002/hed.25356. Epub 2018 Dec 10. PMID 30536465
- [Background] Sugino K, Nagahama M, Kitagawa W, Ohkuwa K, Uruno T, Matsuzu K, Suzuki A, Tomoda C, Hames KY, Akaishi J, Masaki C, Ito K. Risk Stratification of Pediatric Patients with Differentiated Thyroid Cancer: Is Total Thyroidectomy Necessary for Patients at Any Risk? Thyroid. 2020 Apr;30(4):548-556. doi: 10.1089/thy.2019.0231. Epub 2020 Mar 11. PMID 31910105